CLINICAL TRIAL: NCT04814212
Title: Drug-Coated Balloon in Anticoagulated and Bleeding Risk Patients Undergoing PCI
Acronym: DEBATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Collaborators: Central Hospital of Lapland (Unknown); Kuopio University Hospital (Other); Central Finland Hospital District (Other); Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Oulu University Hospital (Other); Tampere University Hospital (Other); Satakunta Central Hospital (Other); Päijät Häme Central Hospital (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Centre Hospitalier de La Rochelle (Other); Hospital Universitario de Cabuenes (Other); University Hospital Carl Gustav Carus (Other); University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Tuomas Rissanen, Head of Heart Center, North Karelia Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEBATE
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: drug-coated balloon; drug eluting stent; coronary artery disease; acute coronary syndrome; percutaneous coronary intervention; DCB; DES; drug coated balloon; drug-eluting stent; drug-eluting balloon; high bleeding risk; HBR
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization to the study groups is done using the Random generator in blocks of 20 without stratification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated balloon (DCB) (Experimental): The coronary lesions fulfilling the inclusion criteria and randomized to the DCB group.
  Interventions: Device: Percutaneous coronary intervention using drug-coated balloon
- Drug-eluting stent (DES) (Active Comparator): The coronary lesions fulfilling the inclusion criteria and randomized to the DES group.
  Interventions: Device: Percutaneous coronary intervention using drug-eluting stent

INTERVENTIONS:
Device: Percutaneous coronary intervention using drug-coated balloon — SeQuent Please (BBraun) + tailored antithrombotic regimen:
  1. Stable patients without OAC: perioperative SAPT (preferably) or perioperative DAPT followed by lifelong SAPT
  2. Stable patients with OAC: perioperative SAPT (preferably) or perioperative DAPT and lifelong OAC
  3. ACS patients without OAC: 1-month DAPT followed by lifelong SAPT
  4. ACS patients with OAC: perioperative DAPT followed by 1-month SAPT and lifelong OAC
  Other Names: DCB
  Arms: Drug-coated balloon (DCB)
Device: Percutaneous coronary intervention using drug-eluting stent — Biofreedom (Biosensors), Synergy (Boston Scientific), Ultimaster Tansei (Terumo) and Integrity Onyx (Medtronic), Xience Pro S (Abbott) or Promus Elite (Boston Scientific) or any other DES can also be used provided that it has a CE mark for 1-month DAPT, combined with tailored antithrombotic regimen:
  1. Stable patients without OAC: 1-month DAPT followed by lifelong SAPT
  2. Stable patients with OAC: perioperative DAPT followed by 6 months SAPT (ADP receptor blocker) and life-long OAC
  3. ACS patients without OAC: 3-month DAPT followed by lifelong SAPT
  4. ACS patients with OAC: perioperative DAPT followed by 6 months SAPT (ADP receptor blocker) and lifelong OAC
  Other Names: DES
  Arms: Drug-eluting stent (DES)

SUMMARY:
The purpose of this study is to compare DCB with DES in stable CAD or ACS patients who are at high risk of bleeding. The hypothesis of the DEBATE trial is that the strategy using DCB and a shorter DAPT regimen is non-inferior to the treatment using DES and longer DAPT duration on patients with high bleeding risk. If non-inferiority is shown, the superiority of the DCB strategy over DES strategy will be tested.

DETAILED DESCRIPTION:
Implantation of a drug-eluting stent (DES) has become a standard of percutaneous coronary intervention (PCI) during the last two decades. However there are still significant drawbacks in using DES as a permanent coronary implant. Most importantly, bleeding remains a significant complication of PCI, especially in elderly patients. The number of PCI patients having OAC:s is already significant, and will grow in the future, as the volume of PCIs in octogenarians increases, and so does the incidence of atrial fibrillation by age. After stenting at least one month lasting dual antiplatlet treatment (DAPT) is mandatory, and it cannot be safely terminated in case of a bleed. The optimal duration of DAPT on patients at bleeding risk is not known.

Balloon coated with paclitaxel and iopromide (drug-coated balloon, DCB) was originally developed for the treatment of in-stent restenosis, but later its potential for the treatment of de-novo coronary artery leasons has become clear in large registry trials. So far, the randomized controlled studies have shown the non-inferiority of PCI using DCB in comparison to DES in de novo leasons in small vessels. Also the non-inferiority of PCI using DCB in comparison to BMS was shown in the DEBUT trial in large vessels on patients at high bleeding risk. These results need to be confirmed in comparison of DCB to DES as the use of BMS is diminishing.

The hypothesis of the DEBATE trial is that the strategy using DCB and a shorter DAPT regimen is non-inferior to the treatment using DES and longer DAPT duration in the treatment of stable CAD or in ACS (UAP or NSTEMI) in patients on anticoagulation medication or otherwise on high bleeding risk. If non-inferiority is shown, the superiority of the DCB strategy over DES strategy will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed written consent
* At least one major or two minor bleeding risk criteria of Academic Research Consortium (ARC)

Major Criteria

* Long-term oral anticoagulation
* Severe or end stage chronic kidney disease (CKD) (estimated glomerular - filtration rate [eGFR] <30 ml/min)
* Hemoglobin <110 g/l
* Spontaneous bleeding requiring hospitalization and transfusion in the past 6 months
* Moderate to severe baseline thrombocytopenia (platelet count <100 x 10e9/L)
* Chronic bleeding diathesis
* Liver cirrhosis with portal hypertension
* Active cancer in the past 12 months
* Previous spontaneous ICH (at any time)
* Previous traumatic ICH within the past 12 months
* Presence of known brain arteriovenous malformation
* Moderate to severe ischemic stroke within the past 6 months
* Nondeferrable major surgery on dual antiplatelet therapy
* Recent major surgery or trauma within 30 days before PCI

Minor Criteria

* Age >75 years
* Moderate CKD (eGFR 30-59 ml/min)
* Hemoglobin 110-129 g/l for men and 110-119 g/l for women
* Spontaneous bleeding requiring hospitalization or transfusion within the past 12 - months not meeting major criterion
* Long term use of oral nonsteroidal antiinflammatory drugs or steroids
* Any ischemic stroke at any time not meeting major criterion

Either of the following:

1. Stabile angina or dyspnea and a coronary narrowing causing myocardial ischemia detected in the angiogram. In stable patients prior PCI, the evidence of ischemia is needed acquired either by perfusion imaging or by pressure wire measurement (FFR) during coronary angiography unless the coronary stenosis is > 90% in diameter.
2. ACS (UAP or NSTEMI): symptoms of heart ischemia≥ 20 minutes and ≥ 0,5mm ST-depression or transient ST-elevation or T-wave inversion at least in two adjacent leads and/or a high sensitivity troponin (hs-tnt) rise at least one unit above the 99. percentil or at least 50% rise in hs-tnt between two samples taken 1-3 hours apart.

At least one of the following:

* ≥1 de novo lesions in native coronary arteries or bypass vein grafts
* Reference diameter of the vessel is 2.0-5.0mm'
* Lesion length ≤ 40mm
* Lesion or lesions are suitable for PCI

Exclusion Criteria:

* Inability to give written consent
* STEMI
* Reference diameter of the vessel is <2.0mm or >5.0 mm
* Bifurcation lesion requiring the stenting of either of the branches after predilatation (TIMI<3 or significant recoil >30% in the main epicardial vessel: LAD, LCX or RCA) after predilatation)
* Dissection affecting the flow (TIMI<3) or significant recoil (>30% in the main epicardial vessel: LAD, LCX or RCA) after predilatation
* in-stent restenosis
* Chronic total occlusion
* Life expectancy < 12 months
* Cardiogenic shock at the arrival to the coronary angiography
* Uncertainty about neurological recovery e.g. after resuscitation
* Need for bypass surgery by heart team decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
The composite of MACE and BARC type 2-5 bleeding episodes | 12 months
  Major Adverse Cardiac Event = a composite of cardiac death, nonfatal myocardial infarction (MI) and ischemia driven-target lesion revascularization (ID-TLR). BARC = Bleeding academic research consortium. In stable patients, the evidence of ischemia is acquired either by non-invasive testing (for example stress ECG or perfusion imaging) or by pressure wire measurement (FFR) during coronary angiography.

SECONDARY OUTCOMES:
The composite of MACE and BARC2-5 bleedings | 24 and 36 months
  Major Adverse Cardiac Event = a composite of cardiac death, nonfatal myocardial infarction (MI) and ischemia driven-target lesion revascularization (ID-TLR). BARC = Bleeding academic research consortium. In stable patients, the evidence of ischemia is acquired either by non-invasive testing (for example stress ECG or perfusion imaging) or by pressure wire measurement (FFR) during coronary angiography.
MACE | 12, 24 and 36 months
  Composite of cardiac death, nonfatal myocardial infarction (MI) and ischemia driven-target lesion revascularization (ID-TLR)
BARC2-5 bleedings | 12, 24 and 36 months
  BARC = Bleeding academic research consortium
BARC3-5 bleedings | 12, 24 and 36 months
  BARC = Bleeding academic research consortium
Total mortality | 12, 24 and 36 months
  All-cause mortality
Cardiovascular mortality | 12, 24 and 36 months
  Cardiovascular death is defined as death resulting from cardiovascular causes. The following categories may be collected:
  1. Death caused by acute MI
  2. Death caused by sudden cardiac, including unwitnessed, death
  3. Death resulting from heart failure
  4. Death caused by stroke
  5. Death caused by cardiovascular procedures
  6. Death resulting from cardiovascular hemorrhage
  7. Death resulting from other cardiovascular cause
TVF | 12, 24 and 36 months
  Target-vessel failure
TLR | 12, 24 and 36 months
  Target-lesion revascularization
TLF | 12, 24 and 36 months
  Target-lesion failure
Myocardial infarction | 12, 24 and 36 months
  Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document will be used (Circulation. 2018;137:2635-2650)
The composite of TVF (Target-vessel failure) and BARC2-5 bleedings | 12, 24 and 36 months
  Target-vessel failure. BARC = Bleeding academic research consortium.
The composite of TLF (Target-lesion failure) and BARC2-5 bleedings | 12, 24 and 36 months
  Target-lesion failure. BARC = Bleeding academic research consortium.
The composite of TLR (Target-lesion revascularization) and BARC2-5 bleedings | 12, 24 and 36 months
  Target-lesion revascularization. BARC = Bleeding academic research consortium.
The composite of TLR (Target-lesion revascularization) and BARC3-5 bleedings | 12, 24 and 36 months
  Target-lesion revascularization. BARC = Bleeding academic research consortium.
Acute vessel closure as defined by the international consensus criteria for definite/probable stent thrombosis | 12, 24 and 36 months
  Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document will be used (Circulation. 2018;137:2635-2650)
Hospitalization for urgent revascularization | 12, 24 and 36 months
  Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document will be used (Circulation. 2018;137:2635-2650)
Stroke (ischemic or hemorrhagic) or TIA | 12, 24 and 36 months
  Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document will be used (Circulation. 2018;137:2635-2650)

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas T Rissanen, MD, PhD, Principal Investigator — North Karelia Central Hospital
Locations (14):
- Finland (10):
  - Central Hospital of Central Finland, Jyväskylä, Central Finland
  - Central Hospital of Lapland, Rovaniemi, Lapland
  - Kuopio University Hospital, Kuopio, Northern Savonia
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki University Hospital, Helsinki, Uusimaa
  - North Karelia Central Hospital, Joensuu
  - Central Hospital of Päijät-Häme, Lahti
  - Oulu university hospital, Oulu
  - Satakunta Central Hospital, Pori
  - Tampere Heart Hospital, Tampere
- Centre Hospitalier La Rochelle, La Rochelle, France
- Germany (2):
  - University Hospital of Carl Gustav Carus, Dresden
  - University Hospital of Saarland, Homburg
- Norfolk and Norwich University Hospital Nhs Foundation Trust, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No